CLINICAL TRIAL: NCT02176421
Title: A Prospective, Open Label Study Evaluating JUVÉDERM® VOLBELLA With Lidocaine Treatment for the Correction of Skin Depressions in the Infra-orbital Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAF-AGN-MED-FIL-020
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Results first posted 2015-07-16 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Infra-orbital Skin Depressions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VOLBELLA® with lidocaine (Experimental): Infra-orbital skin depressions injected with VOLBELLA® with lidocaine.
  Interventions: Device: VOLBELLA® with lidocaine

INTERVENTIONS:
Device: VOLBELLA® with lidocaine — VOLBELLA® with lidocaine administered to correct skin depression during initial treatment and optional top-up treatment 14 days later.

SUMMARY:
A prospective, open label, study evaluating JUVÉDERM® VOLBELLA with lidocaine treatment for the correction of skin depressions in the infra-orbital area (under the eyes)

ELIGIBILITY:
Inclusion Criteria:

* Has Grade > 0 at screening within each eye (bilateral skin depression in the infra-orbital area), as evaluated by the Evaluating Investigator (EI) using AIRS
* Agree to refrain from undergoing other antiwrinkle/volumizing treatments in the upper two-thirds of the face (eyebrow to cheeks/cheekbones) for the duration of the study

Exclusion Criteria:

* Has undergone cosmetic facial procedures [e.g., face-lift, or other surgeries which may alter the appearance of the infra-orbital area (laser, photomodulation, intense pulsed light, radio frequency, dermabrasion, moderate or greater depth chemical peel, or other ablative procedures), tissue augmentation with dermal fillers or fat injections, or mesotherapy] anywhere in the face, or Vistabel® cosmetic injections in the peri-orbital area, within 6 months prior to entry in the study or be planning to undergo any of these procedures at any time during the study. NOTE: Prior treatment with HA fillers and/or collagen is allowed, provided the treatment was administered more than 12 months prior to study entry
* Has undergone volumizing of the mid face within 12 months prior to study entry
* Has ever received semi-permanent fillers or permanent facial implants (e.g., calcium hydroxylapatite, poly-L-lactic acid, polymethylmethacrylate, silicone, expanded polytetrafluoroethylene) anywhere in the infra-orbital area, or be planning to be implanted with any of these products at any time during the study
* Have a history of skin cancer
* Have a history of hypertrophic scarring
* Have a subcutaneous retaining structure on the face (e.g., meshing, gold strand)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-05-15 (Actual); Primary Completion 2014-08-18 (Actual); Study Completion 2015-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Allergan Medical
Locations (1):
- Lyon, Auvergne-Rhône-Alpes, France

REFERENCES:
- [Background] Niforos F, Acquilla R, Ogilvie P, Safa M, Signorini M, Creutz L, Kerson G, Silberberg M. A Prospective, Open-Label Study of Hyaluronic Acid-Based Filler With Lidocaine (VYC-15L) Treatment for the Correction of Infraorbital Skin Depressions. Dermatol Surg. 2017 Oct;43(10):1271-1280. doi: 10.1097/DSS.0000000000001127. PMID 28858926

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VOLBELLA® With Lidocaine
Started | 80
Completed | 75
Not Completed | 5
Not completed — Lost to Follow-up | 4
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | VOLBELLA® With Lidocaine
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.1 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With a ≥1 Grade Improvement From Baseline in Infra-Orbital Area on the Allergan Infra-Orbital Rating Scale (AIRS) on the Right and Left Side
Description: The Investigator evaluated the severity of skin crease and volume loss in the infra-orbital area on both the right and left sides on the 6-point AIRS ranging from 0 (least severe) to 5 (most severe).
Time Frame: Baseline, Month 1
Population: All subjects with data for this outcome measure
Measure: Number; unit: Percentage of Subjects
Arm/Group | VOLBELLA® With Lidocaine
Number analyzed (Participants) | 74
Percentage of Subjects
  Right Side | 99
  Left Side | 100

2. Secondary Outcome: Percentage of Subjects With a ≥1 Grade Improvement From Baseline in Infra-Orbital Area on the AIRS on the Right and Left Side
Description: as for outcome 1
Time Frame: Baseline, Day 0, Day 14, Month 6, Momth 9, Month 12
Population: All subjects with data for this outcome measure
Measure: Number; unit: Percentage of Subjects
Arm/Group | VOLBELLA® With Lidocaine
Number analyzed (Participants) | 76
Percentage of Subjects
  Day 0 Right Side | 99
  Day 0 Left Side | 99
  Day 14 Right Side (N=60) | 98
  Day 14 Left Side (N=60) | 100
  Month 6 Right Side (N=73) | 93
  Month 6 Left Side (N=73) | 92
  Month 9 Right Side (N=72) | 81
  Month 9 Left Side (N=72) | 83
  Month 12 Right Side (N=71) | 55
  Month 12 Left Side (N=71) | 59

3. Secondary Outcome: Injector Ease of Use on an 11-Point Scale
Description: The injectors rated the ease of injection and ease of modeling of the product on an 11-point scale from 0 (extremely difficult) to 10 (extremely easy).
Time Frame: Day 0
Population: All subjects with data for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | VOLBELLA® With Lidocaine
Number analyzed (Participants) | 76
Scores on a Scale | 9.8 (0.0)

4. Secondary Outcome: Percentage of Subjects Assessed by the Investigator as Very Well Improved or Well Improved on the 5-Point Global Aesthetic Improvement Scale (GAIS)
Description: The Investigator evaluated the subjects global aesthetic improvement on right and left sides using the 5-point GAIS (1=Very Well Improved, 2=Well Improved, 3=Improved, 4=Not Improved, 5=Worsened State). The percentage of subjects assessed as Very Well Improved and Well Improved are reported.
Time Frame: Day 0, Day 14, Month 1, Month 6, Month 9, Month 12
Population: All subjects with data for this outcome measure
Measure: Number; unit: Percentage of Subjects
Arm/Group | VOLBELLA® With Lidocaine
Number analyzed (Participants) | 76
Percentage of Subjects
  Day 0 Very Well Improved Right Side | 45
  Day 0 Very Well Improved Left Side | 43
  Day 0 Well Improved Right Side | 34
  Day 0 Well Improved Left Side | 37
  Day 14 Very Well Improved Right Side (N=60) | 68
  Day 14 Very Well Improved Left Side (N=60) | 63
  Day 14 Well Improved Right Side (N=60) | 27
  Day 14 Well Improved Left Side (N=60) | 30
  Month 1 Very Well Improved Right Side (N=76) | 57
  Month 1 Very Well Improved Left Side (N=75) | 65
  Month 1 Well Improved Right Side (N=76) | 38
  Month 1 Well Improved Left Side (N=75) | 31
  Month 6 Very Well Improved Right Side (N=73) | 40
  Month 6 Very Well Improved Left Side (N=73) | 37
  Month 6 Well Improved Right Side (N=73) | 38
  Month 6 Well Improved Left Side (N=73) | 42
  Month 9 Very Well Improved Right Side (N=72) | 18
  Month 9 Very Well Improved Left Side (N=72) | 18
  Month 9 Well Improved Right Side (N=72) | 25
  Month 9 Well Improved Left Side (N=72) | 26
  Month 12 Very Well Improved Right Side (N=71) | 6
  Month 12 Very Well Improved Left Side (N=71) | 6
  Month 12 Well Improved Right Side (N=71) | 23
  Month 12 Well Improved Left Side (N=71) | 27

5. Secondary Outcome: Percentage of Subjects Assessed by the Subjects as Very Well Improved or Well Improved on the 5-Point Global Aesthetic Improvement Scale (GAIS)
Description: The subjects evaluated their global aesthetic improvement on the right and left sides using the 5-point GAIS (1=Very Well Improved, 2=Well Improved, 3=Improved, 4=Not Improved, 5=Worsened State). The percentage of subjects assessed as Very Well Improved and Well Improved are reported.
Time Frame: Day 0, Day 14, Month 1, Month 6, Month 9, Month 12
Population: All subjects with data for this outcome measure
Measure: Number; unit: Percentage of Subjects
Arm/Group | VOLBELLA® With Lidocaine
Number analyzed (Participants) | 76
Percentage of Subjects
  Day 0 Very Well Improved Right Side | 21
  Day 0 Very Well Improved Left Side | 18
  Day 0 Well Improved Right Side | 38
  Day 0 Well Improved Left Side | 36
  Day 14 Very Well Improved Right Side (N=60) | 43
  Day 14 Very Well Improved Left Side (N=60) | 40
  Day 14 Well Improved Right Side (N=60) | 35
  Day 14 Well Improved Left Side (N=60) | 38
  Month 1 Very Well Improved Right Side (N=76) | 39
  Month 1 Very Well Improved Left Side (N=75) | 43
  Month 1 Well Improved Right Side (N=76) | 32
  Month 1 Well Improved Left Side (N=75) | 30
  Month 6 Very Well Improved Right Side (N=73) | 22
  Month 6 Very Well Improved Left Side (N=73) | 18
  Month 6 Well Improved Right Side (N=73) | 29
  Month 6 Well Improved Left Side (N=73) | 30
  Month 9 Very Well Improved Right Side (N=72) | 19
  Month 9 Very Well Improved Left Side (N=72) | 17
  Month 9 Well Improved Right Side (N=72) | 26
  Month 9 Well Improved Left Side (N=72) | 25
  Month 12 Very Well Improved Right Side (N=73) | 16
  Month 12 Very Well Improved Left Side (N=73) | 12
  Month 12 Well Improved Right Side (N=73) | 23
  Month 12 Well Improved Left Side (N=73) | 25

6. Secondary Outcome: Subject Overall Eye Appearance Total Score on the 5-Point Periorbital Aesthetic Appearance Questionnaire (PAAQ)
Description: Subjects assessed their overall eye appearance on the PAAQ. The PAAQ includes 9 questions about how the subject's overall eye appearance affected them over the past 7 days. Each question is assessed on a 5-point scale from 0 (never/best) to 4 (all of the time/worse), with the total score ranging from 0 (best) to 36 (worse).
Time Frame: Day 0, Day 14, Month 1, Month 6, Month 9, Month 12
Population: All subjects with data for this outcome measure
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | VOLBELLA® With Lidocaine
Number analyzed (Participants) | 76
Scores on a Scale
  Day 0 | 19.3 (7.1)
  Day 14 | 7.4 (6.4)
  Month 1 | 6.0 (7.2)
  Month 6 | 9.5 (7.7)
  Month 9 | 9.9 (7.9)
  Month 12 | 10.7 (8.4)

ADVERSE EVENTS:
Time Frame: Adverse event (AE) and serious adverse event (SAE) data were collected for 1 month for each subject. )
Arm/Group | VOLBELLA® With Lidocaine
Serious Adverse Events (participants affected / at risk) | 1/80
Other Adverse Events (participants affected / at risk) | 77/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | VOLBELLA® With Lidocaine (N=80)
Uterine Leiomyoma (Reproductive system and breast disorders) | 1/67 — Females Only
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VOLBELLA® With Lidocaine (N=80)
Injection Site Bruising (General disorders) | 44
Injection Site Erythema (General disorders) | 39
Injection Site Oedema (General disorders) | 32
Injection Site Pain (General disorders) | 26
Injection Site Reaction (General disorders) | 33
Back Pain (Musculoskeletal and connective tissue disorders) | 5
Headache (Nervous system disorders) | 25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.